CLINICAL TRIAL: NCT02054442
Title: A Phase Ib-II Study of the Combination of Cetuximab and Methotrexate in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck. A Study of the Dutch Head and Neck Society
Brief Title: A Study of the Combination of Cetuximab and Methotrexate in Recurrent or Metastatic Cancer of the Head and Neck
Acronym: COMMENCE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Serono International SA (Industry); Leiden University Medical Center (Other); Academisch Ziekenhuis Maastricht (Other); Erasmus Medical Center (Other); Medisch Spectrum Twente (Other); Medical Center Haaglanden (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHN01; 2013-002886-20 (EudraCT Number); DHNS 2013-01 (Other: Dutch Head and Neck Society)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: cetuximab; methotrexate; squamous cell carcinoma head neck; palliative chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: MTX in combination with cetuximab (Experimental): The dosage of cetuximab will be i.v. 400 mg/m2 over a period of 2h for the first infusion, followed by infusions of 250 mg/m2 over 1 hour once weekly. Cetuximab will be dissolved in 500 ml NaCl 0.9%.
  Premedication: H1-receptor antagonist and dexamethasone.
  The dosage of MTX (Methotrexate) will be i.v. 40 mg/m2 once weekly, administered within 5-10 minutes. MTX will be dissolved in 50 ml NaCl 0.9%.
  Premedication: ondansetron 8 mg.
  Treatment will be continued until progressive disease, unacceptable toxicity or refusal by patient.
  Interventions: Drug: Cetuximab; Drug: Methotrexate
- Arm B: MTX (Active Comparator): The dosage of MTX (Methotrexate) will be i.v. 40 mg/m2 once weekly, administered within 5-10 minutes. MTX will be dissolved in 50 ml NaCl 0.9%.
  Premedication: ondansetron 8 mg.
  Treatment will be continued until progressive disease, unacceptable toxicity or refusal by patient.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cetuximab — We will perform a randomized phase II study to investigate in first line if the addition of cetuximab to MTX is beneficial, i.e. improvement in the PFS, for the patient.
  Other Names: Erbitux; L01XC06
  Arms: Arm A: MTX in combination with cetuximab
Drug: Methotrexate
  Other Names: EMTHEXATE; L01BA01

SUMMARY:
The investigators will perform a randomized phase II study to investigate if the addition of cetuximab to MTX is beneficial for the patient. Because no data on this combination are available the investigators will start with a phase Ib study to investigate the feasibility of the schedule.

DETAILED DESCRIPTION:
The addition of cetuximab to cisplatin and 5-FU in recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) showed an improvement of overall survival (OS), progression free survival (PFS) and response rate (RR). However, cisplatin and 5-FU are toxic cytostatics for the vulnerable recurrent or metastatic SCCHN patient. As one of the primary goals in these patients is palliation, in some patients treatment with cisplatin, 5-FU and cetuximab is not feasible owing to a low performance score (PS of 2) or the patient refusal to receive chemotherapy, i.e. cisplatin and 5-FU, possibly influencing quality of life negatively.

Methotrexate is a cytostatic which has shown to have modest activity in recurrent or metastatic SCCHN. The RR is between 14 and 20%, the median PFS is 3 months, and there is no improvement in OS, which is only 6 months. Toxicity of MTX is very low. Patients with a PS of 2 can be treated with MTX. Patients refusing treatment with cisplatin, 5-FU and cetuximab, frequently choose MTX as palliative treatment.

No data are available on the combination of cetuximab and MTX. The investigators will perform a randomized phase II study to investigate if the addition of cetuximab to MTX is beneficial, i.e. an improvement in the PFS, for the patient. Because no data on this combination are available the investigators will start with a phase Ib study to investigate the feasibility of the schedule.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically/histologically-proven SCCHN
* Recurrent or metastatic SCCHN
* At least one measurable lesion as determined by RECIST v1.1 is required. Lesions in previously irradiated areas should not be considered measurable unless there is clear evidence of progression in such lesions since the radiotherapy.
* No prior systemic treatment for recurrent or metastatic disease
* Primary site: (1) oral cavity, (2) oropharynx, (3) hypopharynx, (4) larynx, or (5) unknown primary squamous cell carcinoma in the head and neck region presenting originally with lymph node metastases (N1-N3).
* Time between prior treatment and inclusion in the study (> 3 months). Palliative RT in case of painful bone metastases is allowed in phase II and after 4 weeks in phase Ib
* Ineligible (due to medical co-morbidities) or intolerant to platinum-based therapy per medical history or refusing cisplatin-based chemotherapy by the patient
* WHO performance status 0-2.
* Age >18 years
* Adequate organ function and laboratory parameters as defined by:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109 /L
  * Hemoglobin (Hb) ≥ 9 g/dl 5.6 mmol/l (which may be achieved by transfusion)
  * Platelets (PLT) ≥ 100 x 109/L
  * AST and ALT ≤ 2.5 x ULN (upper limit of normal)
  * Serum bilirubin ≤ 1.5 x ULN
  * Calculated creatinine clearance or MDRD > 60ml/min
* Recovered from all adverse events (AEs) of previous anti-cancer therapies. AEs related to prior radiotherapy are allowed.
* Written informed consent

Exclusion Criteria:

* Serious active infections
* Patients (M/F) with reproductive potential not implementing adequate contraceptives measures
* Prior treatment with EGFR inhibitors or MTX
* Concomitant (or within 4 weeks before randomization) administration of any other experimental drug under investigation
* Concurrent treatment with any other anti-cancer therapy.
* Central nervous system involvement
* Lung fibrosis
* Pleural effusion or ascites or other third space effusions
* History of another malignancy within 2 years prior to starting study treatment, except cured basal cell carcinoma of the skin, excised carcinoma in situ of the cervix, or other head and neck cancer.
* Pregnancy or lactation
* Any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, social/psychological complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-08; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | During the first 4 weeks after start of the combination MTX and cetuximab
  In the phase Ib study: toxicity scored with CTC v 4.0*; incidence of dose limiting toxicity (DLT) during the first 4 weeks after start of the combination
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  In the phase II study: progression free survival (PFS). The analysis of PFS can be performed as soon as the target event (progression or death) has been observed in 98 of the 114 subjects randomized.

SECONDARY OUTCOMES:
Overall survival (OS) | Followed up to 12 months after randomization
  Overall survival (OS) The analysis of OS can be performed as soon as the target event has been observed in 98 of the 114 subjects randomized.
Response rate (RR) | Till end of treatment
  The difference in RR rates between both treatment arms will be analyzed using a stratified Cochran Mantel Haenszel test at a one-sided alpha-level of 0.05. In addition to the response rates in both arms, the odds ratio will be reported together with 90% confidence intervals. The impact of various demographic and disease characteristics (e.g. HPV positivity), on RR will be investigated using an exploratory logistic regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Carla M van Herpen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (8):
- Netherlands (8):
  - Medisch Spectrum Twente, Enschede
  - Medical Centre Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud university medical center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Medical Centre Haaglanden, The Hague
  - St. Elisabeth Ziekenhuis, Tilburg